CLINICAL TRIAL: NCT02161263
Title: Patient Quality of Vision and Quality of Life With LASIK Surgery
Brief Title: Quality of Vision and Quality of Life With LASIK
Status: Completed | Type: Observational
Sponsor: Edward E. Manche (Other)
Responsible Party: Sponsor-Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 30301
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Myopia; Astigmatism; Quality of Lifte
Keywords: LASIK; Satisfaction
MeSH Terms: conditions — Myopia; Astigmatism; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of Vision after LASIK surgery: Questionnaire
  Interventions: Other: Patient Quality of Life andVision after LASIK Surgery

INTERVENTIONS:
Other: Patient Quality of Life andVision after LASIK Surgery — Patient questionnaire

SUMMARY:
The investigators are administering a validated questionnaire looking at patient reported quality of life and quality of vision after LASIK surgery

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the prevalence of any functional limitations and their associated factors at one, three, six, and twelve months after LASIK surgery and finally the level of patient satisfaction, including the prevalence of any dissatisfaction and its associated factors at one, three, six and twelve months following LASIK surgery using two questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 21 years or older.
* Have the ability to give informed consent.
* Speak and read English fluently.
* Have not previously had any form of refractive surgery, including prior LASIK or cataract surgery.
* May benefit from increased spectacle independence.
* Have been determined to be a good candidate for the LASIK procedure based on the investigator's assessment of medical and ophthalmic health, general cognitive function, and physical and social limitations.
* Have a treatment target of bilateral emmetropia.
* Express willingness and potential ability to return for all follow-up examinations through the 12-month follow-up exam under the care of the treating investigator.
* Are not enrolled in any other research study.

Exclusion Criteria:

* Subjects under the age of 21.
* Patients with excessively thin corneas.
* Patients with topographic evidence of keratoconus.
* Patients with ectactic eye disorders.
* Patients with autoimmune diseases.
* Patients who are pregnant or nursing.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 21 with healthy eyes and nearsightedness, farsightedness and/or astigmatism
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Quality of Vision and Quality of Life Questionnaires after LASIK Surgery | 12 months
  Patients will complete questionnaires preoperatively and postoperatively at month twelve.

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Eye Laser Center, Palo Alto, California, United States